CLINICAL TRIAL: NCT04490707
Title: Clinical Study of Azacytidine Combined With Lenalidomide As Maintenance Therapy Based on MRD Monitoring In Elderly or Unfit Patients With Acute Myeloid Leukemia
Brief Title: Study of Azacytidine Combined With Lenalidomide As Maintenance Therapy Based on MRD Monitoring in AML
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ge Zheng (Other)
Responsible Party: Sponsor-Investigator, Ge Zheng, Director of Department of Hematology, Zhongda Hospital
Organization: Zhongda Hospital (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZDYYGZ202005
Record Dates: First submitted 2020-07-26; First posted 2020-07-29 (Actual); Last update posted 2022-03-24 (Actual); Status verified 2022-03

CONDITIONS: Acute Myeloid Leukemia in Remission
Keywords: Acute myeloid leukemia; Azacitidine; Lenalidomide; Maintenance Therapy; MRD
MeSH Terms: conditions — Leukemia, Myeloid, Acute | interventions — Azacitidine; Lenalidomide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Azacitidine plus Lenalidomide (AZA+LEN) (Experimental): Arm 1(AZA+LEN): Elderly or unfit for intensive therapy AML patients who had achieved CR after remission-induction and consolidation chemotherapy enter maintenance therapy with AZA combined with LEN: AZA 50mg/m² per day for days 1-5 and LEN 10mg per day orally for days 6-26 , every 28 days for up to 12 cycles or progression.
  AZA -Azacitidine, LEN- Lenalidomide
  Interventions: Drug: Azacitidine; Drug: Lenalidomide
- Azacitidine(AZA) (Experimental): Arm 2 (AZA): Elderly or unfit for intensive therapy AML patients who had achieved CR after remission-induction and consolidation chemotherapy enter maintenance therapy with AZA 50mg/m² per day for days 1-5, every 28 days for up to 12 cycles or progression.
  AZA -Azacitidine
  Interventions: Drug: Azacitidine
- Observation (No Intervention): Arm 3(Observation): Elderly or unfit for intensive therapy AML patients who had achieved CR after remission-induction and consolidation chemotherapy enter observation.

INTERVENTIONS:
Drug: Azacitidine — Elderly or unfit for intensive therapy patients with acute myeloid leukemia who had entered CR receive maintenance therapy contained Azacitidine
  Other Names: AZA
  Arms: Azacitidine plus Lenalidomide (AZA+LEN); Azacitidine(AZA)
Drug: Lenalidomide — Elderly or unfit for intensive therapy patients with acute myeloid leukemia who had entered CR receive maintenance therapy contained Lenalidomide
  Other Names: LEN
  Arms: Azacitidine plus Lenalidomide (AZA+LEN)

SUMMARY:
Great progress has been witnessed on the treatment of acute myeloid leukemia (AML) in recent years. However, elderly patients ineligible for receiving high dose chemotherapy and allo-HSCT, have high relapse rate and treatment-related complications. Azacitidine (AZA), a listed hypomethylating agent in China in 2018, is the only approved demethylating drug in the treatment of AML, following the NCCN guidelines. In addition, lenalidomide(LEN) has been shown to rapidly enhance cytotoxic T- and natural killer (NK)-cell function and reduce relapse post-chemotherapy in patients with MM, also has substantial activity as a single agent in elderly patients with AML. Measurable residual disease (MRD) has been proven to be highly prognostic in quite a number clinical studies. This study is aimed to validate the efficacy and safety advantages of the maintenance therapy that contain AZA and LEN in elderly or unfit for intensive therapy patients with AML based on MRD monitoring.

DETAILED DESCRIPTION:
In this study, elderly or unfit for intensive therapy AML patients who had achieved complete remission(CR) after remission-induction and consolidation chemotherapy were assigned to 3 Arms: (1) Maintenance therapy with AZA combined with LEN（AZA+LEN）: AZA 50mg/m² per day for days 1-5 and LEN 10mg per day orally for days 6-26 , every 28 days for up to 12 cycles or progression; (2) Maintenance therapy with AZA only: AZA 50mg/m² per day for days 1-5, every 28 days for up to 12 cycles or progression; (3) Observation or with supporting therapy. MRD will be assessed by flow cytometry and molecular techniques. The efficacy and safety of the 3 Arms will be evaluated in this study.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with acute myeloid leukemia.Meet the criteria of the 2016 WHO classification system(APL were excluded), based on morphology, immunology, cytogenetics and molecular biology (MICM) diagnosis.
* Complete remission was evaluated according to 2020 NCCN guidelines after induction treatment.
* Patients with age≥ 60 years; or age<60 years unfit for intensive chemotherapy.
* Volunteered to sign the informed consent.

Exclusion Criteria:

* Mental disorders or other conditions that cannot meet the requirements of research, treatment and monitoring.
* Allergic to Azacytidine, Lenalidomide , or other drugs of this study
* Age over 80 years.
* Any other conditions considered by the study investigators that are not suitable for participating in this clinical trial.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Estimated)
Dates: Start 2020-09-01 (Actual); Primary Completion 2022-12-30 (Estimated); Study Completion 2022-12-30 (Estimated)

PRIMARY OUTCOMES:
DFS | From date of randomization or complete remission until the date of first documented disease progression from any cause,assessed up to 100weeks
  DFS in months, in present of disease free survival period of all participants
OS | From date of randomization until the date of first documented death from any cause or end of this study, whichever come first,assessed up to 100weeks
  OS in months, in present of over all survival period of all participants

SECONDARY OUTCOMES:
Adverse events rates | From date of randomization or initial treatment until the end date of the study, assessed up to 100 weeks
  Adverse events rates in percentage

CONTACTS AND LOCATIONS:
Overall Officials: Zheng Ge, M.D, Ph.D, Study Director — Zhongda Hospital
Locations (1):
- Department of Hematology, Zhongda Hospital Southeast University, Institute of Hematology Southeast University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No